CLINICAL TRIAL: NCT04406714
Title: Scaling Colorectal Cancer Screening Through Outreach, Referral, and Engagement (SCORE): A State-Level Program to Reduce Colorectal Cancer Burden in Vulnerable Populations
Brief Title: Scaling CRC Screening Through Outreach, Referral, and Engagement (SCORE)
Acronym: SCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LCCC2056; 4UH3CA233251-02 (NIH)
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer
Keywords: Cancer Screening; Colonoscopy; Community Health Centers; Implementation Science; Patient Navigation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Trial (Age Group 50-75) Using a randomized controlled trial study design, subjects are assigned to one of two arms: Arm 1: Trial Mailed FIT Intervention; or Arm 2: Trial Usual Care. Arm 1 (intervention) receives a mailed FIT plus up to two reminder letters. Subjects are randomized 1:1 at baseline and remain in their assigned arm for the duration of the study (i.e., two annual rounds of mailed FIT).
  Sub-study (Age Group 45-49) Subjects, ages 45-49, are randomly assigned to one of two arms: Arm 3: Sub-Study Mailed FIT Intervention - Enhanced Envelope; or Arm 4: Sub-study Mailed FIT Active Comparator Plain Envelope. Subjects in both Arm 3 and Arm 4 receive mailed FIT plus up to two reminder letters. Subjects are randomized 1:1 at baseline and remain in their assigned arm for the duration of the sub-study (i.e., one annual round of mailed FIT).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Trial Mailed FIT Intervention - Age Group 50-75 (Experimental): Subjects randomized to this arm are 50-75 years of age and eligible for CRC screening using FIT per electronic health record at either of two FQHCs. Only subjects who are 50-75 years of age are randomized to this arm. Subjects who are 50-75 cannot be randomized to Arm 3 or Arm 4.
  Interventions: Behavioral: Trial Mailed FIT Intervention - Age Group 50-75
- Trial Usual Care - Age Group 50-75 (No Intervention): Subjects randomized to this arm are 50-75 years of age and eligible for CRC screening using FIT per electronic health record at either of two FQHCs. Only subjects who are 50-75 years of age are randomized to this arm. Subjects who are 50-75 cannot be randomized to Arm 3 or Arm 4.
- Sub-study Mailed FIT Intervention Enhanced Envelope - Age Group 45-49 (Experimental): Subjects randomized to this arm are 45-49 years of age and eligible for CRC screening using FIT per electronic health record at one FQHC. Only subjects who are 45-49 years of age are randomized to this arm. Subjects who are 45-49 years of age cannot be randomized to Arm 1 or Arm 2 of the main trial.
  Interventions: Behavioral: Sub-Study Mailed FIT Intervention Enhanced Envelope - Age Group 45-49
- Sub-study Mailed FIT Comparator Plain Envelope - Age Group 45-49 (Active Comparator): Subjects randomized to this arm are 45-49 years of age and eligible for CRC screening using FIT per electronic health record at one FQHC. Only subjects who are 45-49 years of age are randomized to this arm. Subjects who are 45-49 years of age cannot be randomized to Arm 1 or Arm 2 of the main trial.
  Interventions: Behavioral: Sub-Study Mailed FIT Active Comparator Plain Envelope - Age Group 45-49

INTERVENTIONS:
Behavioral: Trial Mailed FIT Intervention - Age Group 50-75 — Subjects are mailed an introductory letter advising them that they will receive a FIT kit in the mail. Next, subjects are mailed a FIT packet in an envelope that contains a cover letter, CRC information sheet, FIT instruction sheet, and FIT kit with a pre-paid return envelope. Subjects receive up to two mailed letters reminding them to complete and return the FIT. Subjects receive FIT results via letter or phone call.
  Arms: Trial Mailed FIT Intervention - Age Group 50-75
Behavioral: Sub-Study Mailed FIT Intervention Enhanced Envelope - Age Group 45-49 — Subjects are mailed an introductory letter advising them that they will receive a FIT kit in the mail. Next, subjects are mailed a FIT packet in an enhanced envelope that contains a cover letter, CRC information sheet, FIT instruction sheet, and FIT kit with a pre-paid return envelope. The enhanced envelope is a yellow padded envelope with a USPS tracking label and sticker message: "Important information from your doctor". Subjects receive up to two mailed letters reminding them to complete and return the FIT. Subjects receive FIT results via letter or phone call.
  Arms: Sub-study Mailed FIT Intervention Enhanced Envelope - Age Group 45-49
Behavioral: Sub-Study Mailed FIT Active Comparator Plain Envelope - Age Group 45-49 — Subjects are mailed an introductory letter advising them that they will receive a FIT kit in the mail. Next, subjects are mailed a FIT packet in plain envelope that contains a cover letter, CRC information sheet, FIT instruction sheet, and FIT kit with a pre-paid return envelope. The plain envelope is a white envelope without a USPS tracking label or sticker message. Subjects receive up to two mailed letters reminding them to complete and return the FIT. Subjects receive FIT results via letter or phone call.
  Arms: Sub-study Mailed FIT Comparator Plain Envelope - Age Group 45-49

SUMMARY:
This study will test the effectiveness of mailing fecal immunochemical tests (FITs) in increasing colorectal cancer (CRC) screening rates in U.S. adults ages 45-75. We are implementing this study in two age groups, 45-49 years and 50-75 years.

DETAILED DESCRIPTION:
Trial (Age Group 50-75) This randomized controlled trial assesses the effectiveness, feasibility, acceptability, and cost-effectiveness of mailing FITs from a central location to patients served by FQHCs. Subjects are randomly selected and assigned to receive either a mailed FIT intervention (Arm 1: Trial Mailed FIT Intervention - Age Group 50-75) or usual care (Arm 2: Trial Usual Care - Age Group 50-75). To assess United States Preventive Services Task Force recommendations for annual screening, we will mail subjects one round of FIT per year for up to two years.

Sub-study (Age Group 45-49) A sub-study assesses the effectiveness of mailing FITs from a central location to patients who are 45-49 years of age and newly eligible for CRC screening. The sub-study also assesses the impact of varying the appearance of the FIT packet mailing envelope on FIT return. All eligible patients from one FQHC clinic site are randomly assigned to receive either a mailed FIT intervention that includes an enhanced mailing envelope (Arm 3: Sub-study Mailed FIT Intervention Enhanced Envelope - Age Group 45-49) or a plain envelope (Arm 4: Sub-study Mailed FIT Active Comparator Plain Envelope - Age Group 45-49).

The Trial (Age Group 50-75) and the Sub-study (Age Group 45-49) also assess the effectiveness of delivering patient navigation from a central location to facilitate follow up colonoscopy for patients with a positive (abnormal) FIT result.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 years
* At average risk for CRC ("average risk" is defined as those patients who do not have any of the following: documented history of CRC, colorectal neoplasms, colorectal polyps, colonic adenomas, family history of CRC among first degree relative [father, mother, sister, brother], or diagnosis of inflammatory bowel disease)
* No record of fecal occult blood test (FOBT)/FIT within the past 12 months or colonoscopy within 10 years, sigmoidoscopy within 5 years, barium enema within 5 years, or computed tomography (CT) colonography within 10 years of the EHR query date
* No record of any CRC diagnosis or total colectomy
* No record of comorbidities or screening contraindications, including dementia, hospice care, assisted living, end-stage renal disease, and other cancers (glioblastoma, pancreatic cancer, lung cancer, esophageal cancer, liver and bile duct cancer, mesothelioma)
* Has a complete North Carolina mailing address in the EHR
* Active patient of the clinic (seen within the past 18 months) at the time of randomization
* No record of a positive (abnormal) FIT result in the first study round (Trial Ages 50-75 only)

Exclusion Criteria:

* Age younger than 45 years or older than 75 years
* Not at average risk for CRC ("average risk" is defined as those patients who do not have any of the following: documented history of CRC, colorectal neoplasms, colorectal polyps, colonic adenomas, family history of CRC among first degree relative [father, mother, sister, brother], or diagnosis of inflammatory bowel disease)
* Record of FOBT/FIT within the past 12 months or colonoscopy within 10 years, sigmoidoscopy within 5 years, barium enema within 5 years, or CT colonography within 10 years of the EHR query date
* Record of any CRC diagnosis or total colectomy
* Record of comorbidities or screening contraindications, including dementia, hospice care, assisted living, end-stage renal disease, and other cancers (glioblastoma, pancreatic cancer, lung cancer, esophageal cancer, liver and bile duct cancer, mesothelioma)
* Does not have a complete North Carolina mailing address in the EHR
* Not an active patient of the clinic (not seen within the past 18 months) at the time of randomization
* Record of a positive (abnormal) FIT result reported during the first study round (Trial Ages 50-75)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4318 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reuland, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Roanoke Chowan Community Health Center, Ahoskie, North Carolina
  - Blue Ridge Health, Hendersonville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
As outlined in the Notice of Award, each study site must make its Limited Data Set (LDS) accessible to other sites in the ACCSIS consortium. Information Management Services (IMS) will serve as the repository and have responsibility for creating a Limited Consolidated Data Set (LCDS) for analytic use of researchers both within and external to the ACCSIS consortium. Dataset Items in the LDS are defined by the Common Data Elements. There also will be a "public use data set" that consists of the Common Data Elements, available to external researchers. IMS will use a systematic process to remove identifiers. In addition, all data that underlie results in publications will be available per Cancer Moonshot Notice of Award.
Supporting Information: Study Protocol
Time Frame: The IPD sharing time frame has not been defined at this time.
Access Criteria: There are 2 classes of dataset requests: public use and special. Requests are submitted via the IMS website. Requestors electronically sign and submit necessary forms, including an agreement to acknowledge ACCSIS in publications and presentations. A public use dataset containing common data elements is made available to external researchers by application. IMS responds to public use dataset applications by sending the requestor one-time access to a data download link. External researchers may also request a more customized data set. Requestors must submit a brief concept form or ancillary studies form, for preliminary review by the ACCSIS Steering Committee (SC), before invitation to submit a full proposal. Full proposals receive administrative review by NCI and RTI before being sent to the SC for review and approval. Requestors report every 6 months and published articles or conference presentations to RTI. Requestors are encouraged to make articles available through PubMed Central.

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: colorectal cancer screening test use--United States, 2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 8;62(44):881-8. PMID 24196665
- [Background] Church TR, Yeazel MW, Jones RM, Kochevar LK, Watt GD, Mongin SJ, Cordes JE, Engelhard D. A randomized trial of direct mailing of fecal occult blood tests to increase colorectal cancer screening. J Natl Cancer Inst. 2004 May 19;96(10):770-80. doi: 10.1093/jnci/djh134. PMID 15150305
- [Background] Daly JM, Levy BT, Merchant ML, Wilbur J. Mailed fecal-immunochemical test for colon cancer screening. J Community Health. 2010 Jun;35(3):235-9. doi: 10.1007/s10900-010-9227-8. PMID 20127156
- [Background] Gupta S, Halm EA, Rockey DC, Hammons M, Koch M, Carter E, Valdez L, Tong L, Ahn C, Kashner M, Argenbright K, Tiro J, Geng Z, Pruitt S, Skinner CS. Comparative effectiveness of fecal immunochemical test outreach, colonoscopy outreach, and usual care for boosting colorectal cancer screening among the underserved: a randomized clinical trial. JAMA Intern Med. 2013 Oct 14;173(18):1725-32. doi: 10.1001/jamainternmed.2013.9294. PMID 23921906
- [Background] Jonas DE, Russell LB, Sandler RS, Chou J, Pignone M. Value of patient time invested in the colonoscopy screening process: time requirements for colonoscopy study. Med Decis Making. 2008 Jan-Feb;28(1):56-65. doi: 10.1177/0272989X07309643. PMID 18263561
- [Background] Kempe KL, Shetterly SM, France EK, Levin TR. Automated phone and mail population outreach to promote colorectal cancer screening. Am J Manag Care. 2012 Jul;18(7):370-8. PMID 22823531
- [Background] Levy BT, Daly JM, Xu Y, Ely JW. Mailed fecal immunochemical tests plus educational materials to improve colon cancer screening rates in Iowa Research Network (IRENE) practices. J Am Board Fam Med. 2012 Jan-Feb;25(1):73-82. doi: 10.3122/jabfm.2012.01.110055. PMID 22218627
- [Background] Sabatino SA, Lawrence B, Elder R, Mercer SL, Wilson KM, DeVinney B, Melillo S, Carvalho M, Taplin S, Bastani R, Rimer BK, Vernon SW, Melvin CL, Taylor V, Fernandez M, Glanz K; Community Preventive Services Task Force. Effectiveness of interventions to increase screening for breast, cervical, and colorectal cancers: nine updated systematic reviews for the guide to community preventive services. Am J Prev Med. 2012 Jul;43(1):97-118. doi: 10.1016/j.amepre.2012.04.009. PMID 22704754
- [Background] Siegel RL, Sahar L, Robbins A, Jemal A. Where can colorectal cancer screening interventions have the most impact? Cancer Epidemiol Biomarkers Prev. 2015 Aug;24(8):1151-6. doi: 10.1158/1055-9965.EPI-15-0082. Epub 2015 Jul 8. PMID 26156973
- [Background] US Preventive Services Task Force; Bibbins-Domingo K, Grossman DC, Curry SJ, Davidson KW, Epling JW Jr, Garcia FAR, Gillman MW, Harper DM, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Owens DK, Phillips WR, Phipps MG, Pignone MP, Siu AL. Screening for Colorectal Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2016 Jun 21;315(23):2564-2575. doi: 10.1001/jama.2016.5989. PMID 27304597
- [Derived] Ganguly AP, O'Leary MC, Crockett SD, Ferrari RM, Randolph CM, Stradtman LR, Moore AA, Su K, Tan X, Brenner AT, Reuland DS. Time to Follow-Up Colonoscopy After Positive Fecal Immunochemical Test with Centralized Patient Navigation: A Randomized Clinical Trial. J Gen Intern Med. 2026 Feb 4. doi: 10.1007/s11606-025-10151-2. Online ahead of print. PMID 41639370
- [Derived] Ferrari RM, Randolph CM, O'Leary MC, Lich KH, Moore AA, Leeman J, Brenner AT, Wheeler SB, Crockett SD, Reuland DS. What makes patient navigation work? Identifying functions and forms and conducting causal loop diagramming to specify components of a successful colorectal cancer patient navigation program. Implement Sci Commun. 2026 Jan 19. doi: 10.1186/s43058-026-00858-6. Online ahead of print. PMID 41549310
- [Derived] Reuland DS, O'Leary MC, Crockett SD, Farr DE, Ferrari RM, Malo TL, Moore AA, Randolph CM, Ratner S, Stradtman LR, Stylianou C, Su K, Tan X, Tang V, Wheeler SB, Brenner AT. Centralized Colorectal Cancer Screening Outreach in Federally Qualified Health Centers: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2446693. doi: 10.1001/jamanetworkopen.2024.46693. PMID 39585696
- [Derived] O'Leary MC, Reuland DS, Correa SY, Moore AA, Malo TL, Tan X, Rohweder CL, Wheeler SB, Brenner AT. Uptake of colorectal cancer screening after mailed fecal immunochemical test (FIT) outreach in a newly eligible 45-49-year-old community health center population. Cancer Causes Control. 2023 Dec;34(Suppl 1):125-133. doi: 10.1007/s10552-023-01717-8. Epub 2023 Jun 10. PMID 37300632
- [Derived] Malo TL, Correa SY, Moore AA, Ferrari RM, Leeman J, Brenner AT, Wheeler SB, Tan X, Reuland DS; Scaling Colorectal Cancer Screening Through Outreach, Referral, and Engagement (SCORE) Study Protocol Consortium. Centralized colorectal cancer screening outreach and patient navigation for vulnerable populations in North Carolina: study protocol for the SCORE randomized controlled trial. Implement Sci Commun. 2021 Oct 7;2(1):113. doi: 10.1186/s43058-021-00194-x. PMID 34620250
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — https://unclineberger.org/patientcare/clinical-trials/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were enrolled between 07/07/2020 - 02/28/2022 in one center in North Carolina.
Groups:
- Experimental: Trial Mailed FIT - Age Group 50-75: Subjects randomized to this arm are 50-75 years of age and eligible for CRC screening using FIT per electronic health record at either of the two study sites. This arm receives a mailed FIT and up to two reminder letters.
- No Intervention: Trial Usual Care - Age Group 50-75: Subjects randomized to this arm are 50-75 years of age and eligible for CRC screening using FIT per electronic health record at either of the two study sites. This arm receives the usual care.
- Experimental: Sub-study Mailed FIT Age Group 45-49 Enhanced Envelope: Subjects randomized to this arm are 45-49 years of age and eligible for CRC screening using FIT per electronic health record at one study site. This arm receives a mailed FIT in an enhanced mailing envelope and up to two reminder letters.
- Active Comparator: Sub-study Mailed FIT Comparator Plain Envelope - Age Group 45-49: Subjects randomized to this arm are 45-49 years of age and eligible for CRC screening using FIT per electronic health record at one study site. This arm receives a mailed FIT in a plain envelope and up to two reminder letters.
Period: Overall Study
Arm/Group | Experimental: Trial Mailed FIT - Age Group 50-75 | No Intervention: Trial Usual Care - Age Group 50-75 | Experimental: Sub-study Mailed FIT Age Group 45-49 Enhanced Envelope | Active Comparator: Sub-study Mailed FIT Comparator Plain Envelope - Age Group 45-49
Started | 2001 | 2001 | 158 | 158
Completed | 2001 | 2001 | 158 | 158
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Trial Mailed FIT - Age Group 50-75 | No Intervention: Trial Usual Care - Age Group 50-75 | Experimental: Sub-study Mailed FIT Age Group 45-49 Enhanced Envelope | Active Comparator: Sub-study Mailed FIT Comparator Plain Envelope - Age Group 45-49 | Total
Number analyzed (Participants) | 2001 | 2001 | 158 | 158 | 4318
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1487 | 1496 | 158 | 158 | 3299
  >=65 years | 514 | 505 | 0 | 0 | 1019
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1135 | 1121 | 84 | 97 | 2437
  Male | 866 | 880 | 74 | 61 | 1881
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 185 | 179 | 13 | 12 | 389
  Not Hispanic or Latino | 1687 | 1679 | 141 | 145 | 3652
  Unknown or Not Reported | 129 | 143 | 4 | 1 | 277
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 8 | 1 | 2 | 15
  Asian | 17 | 10 | 0 | 3 | 30
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 1 | 0 | 5
  Black or African American | 549 | 536 | 88 | 96 | 1269
  White | 1272 | 1295 | 50 | 44 | 2661
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 156 | 151 | 18 | 13 | 338
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2001 | 2001 | 158 | 158 | 4318

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Completed Colorectal Cancer (CRC) Screening Within 6 Months (Trial - Age Group 50-75)
Description: "The proportion of subjects who received study Intervention (Age Group 50-75) and did not receive study intervention (Usual Care - Age Group 50-75 who completed CRC screening using any of the screening modalities recommended by the United States Preventive Services Task Force per electronic health record review.
  Fecal immunochemical test (FIT), fecal occult blood test [FOBT], fecal immunochemical test - deoxyribonucleic acid (FIT-DNA), colonoscopy, flexible sigmoidoscopy, flexible sigmoidoscopy with FIT, Computerized Tomography colonography."
Time Frame: Up to 6 months after randomization
Population: Subjects who actively receive health care from the study sites, aged between 50-75.
Measure: Count of Participants; unit: Participants
Groups:
- Trial Mailed FIT Intervention - Age Group 50-75: Subjects who are between 50-75 years of age and received study intervention.
  Trial Mailed FIT Intervention: Subjects are mailed an introductory letter advising them that they will receive a FIT kit in the mail. Next, subjects are mailed a FIT packet in an envelope that contains a cover letter, CRC information sheet, FIT instruction sheet, and FIT kit with a pre-paid return envelope. Subjects receive up to two mailed letters reminding them to complete and return the FIT. Subjects receive FIT results via letter or phone call.
- Trial Usual Care - Age Group 50-75: Subjects who are 50-75 years of age and did not receive study intervention.
Arm/Group | Trial Mailed FIT Intervention - Age Group 50-75 | Trial Usual Care - Age Group 50-75
Number analyzed (Participants) | 2001 | 2001
Participants | 598 | 192

2. Secondary Outcome: Proportion of Subjects Who Returned a Completed Mailed FIT at 60 Days
Description: The proportion of subjects who received study Intervention (Age Group - 50-75) and returned a completed FIT per electronic health record review.
Time Frame: Up to 60 days after randomization
Population: Subjects who actively receive health care from the study sites, aged between 50-75.
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Mailed FIT Intervention - Age Group 50-75
Number analyzed (Participants) | 2001
Participants | 409

3. Secondary Outcome: Proportion of Subjects Who Completed a Follow-up (Diagnostic) Colonoscopy
Description: The proportion of subjects who received study Intervention (Age Group 50-75) and did not receive study information (Usual Care only - Age Group 50-75), who had a positive (abnormal) FIT/FOBT result, and for whom colonoscopy was deemed to be clinically appropriate by the subject's provider, who completed follow-up (diagnostic) colonoscopy per electronic health record review.
Time Frame: Up to 6 months after diagnostic colonoscopy referral date
Population: Subjects who started the study and were assessed for colon carcinoma within 6 months.
Measure: Count of Participants; unit: Participants
Groups:
- Trial Mailed FIT Intervention - Age Group 50-75: Subjects are 50-75 years of age and eligible for CRC screening using FIT per electronic health record at either of the two study sites. Subjects with an abnormal FIT result following randomization and receipt of the mailed FIT intervention are offered navigation support, in addition to usual care, to complete diagnostic colonoscopy
  Trial Mailed FIT Intervention: Subjects are mailed an introductory letter advising them that they will receive a FIT kit in the mail. Next, subjects are mailed a FIT packet in an envelope that contains a cover letter, CRC information sheet, FIT instruction sheet, and FIT kit with a pre-paid return envelope. Subjects receive up to two mailed letters reminding them to complete and return the FIT. Subjects receive FIT results via letter or phone call.
- Trial Usual Care - Age Group 50-75: Subjects are 50-75 years of age and eligible for CRC screening using FIT per electronic health record at either of the two study sites. Subjects with an abnormal FIT result following randomization to this arm receive usual care only to complete diagnostic colonoscopy.
Arm/Group | Trial Mailed FIT Intervention - Age Group 50-75 | Trial Usual Care - Age Group 50-75
Number analyzed (Participants) | 81 | 26
Participants
  Abnormal FIT | 48 | 18
  Completed colonoscopy | 33 | 8

4. Secondary Outcome: Number of Subject Colorectal Carcinoma (CRC) and Advanced Adenomas Detected at 12 Months
Description: Number of CRCs and advanced adenomas detected among subjects who received study Intervention (Age Group 50-75) and subjects who did not receive study intervention (Usual Care only - Age Group 50-75) per electronic health record review.
Time Frame: Up to 12 months after screening or diagnostic colonoscopy result date
Population: Subjects who participated to the study and were diagnosed with colorectal carcinoma.
Measure: Count of Participants; unit: Participants
Groups:
- Trial Mailed FIT Intervention - Age Group 50-75: Subjects randomized to this arm are 50-75 years of age and eligible for CRC screening using FIT per electronic health record at either of the two study sites. Only subjects who are 50-75 years of age are randomized to this arm.
  Trial Mailed FIT Intervention - Age Group 50-75: Subjects are mailed an introductory letter advising them that they will receive a FIT kit in the mail. Next, subjects are mailed a FIT packet in an envelope that contains a cover letter, CRC information sheet, FIT instruction sheet, and FIT kit with a pre-paid return envelope. Subjects receive up to two mailed letters reminding them to complete and return the FIT. Subjects receive FIT results via letter or phone call.
- Trial Usual Care - Age Group 50-75: Subjects randomized to this arm are 50-75 years of age and eligible for CRC screening using FIT per electronic health record at either of the two study sites. Only subjects who are 50-75 years of age are randomized to this arm.
Arm/Group | Trial Mailed FIT Intervention - Age Group 50-75 | Trial Usual Care - Age Group 50-75
Number analyzed (Participants) | 598 | 192
Participants | 22 | 8

5. Secondary Outcome: Number of Days From CRC Diagnosis to the Date of Evaluation for CRC Treatment
Description: Number of days from CRC diagnosis to the date of evaluation for CRC treatment among subjects who received study Intervention (Age Group 50-75) and subjects who did not receive study intervention (Usual Care - Age Group 50-75) using electronic health record data to ascertain the dates of CRC diagnosis and evaluation for CRC treatment.
Time Frame: Up to 12 months after CRC diagnosis
Population: Participants were diagnosed with CRC ever during Round 1. Five subjects from Trial Mailed FIT Intervention - Age Group 50-75 and 2 subjects from Trial Usual Care - Age Group 50-75 were evaluated for treatment.
Measure: Mean (Full Range); unit: days
Arm/Group | Trial Mailed FIT Intervention - Age Group 50-75 | Trial Usual Care - Age Group 50-75
Number analyzed (Participants) | 5 | 2
days | 3.25 [0 to 13] | 0 [0 to 0]

6. Secondary Outcome: Number of Subjects Who Received Referral for Cancer Treatment
Description: Number of subjects who received study Intervention (Age Group 50-75) and did not receive intervention (Age Group 50-75) who received referral for cancer treatment among individuals diagnosed with CRC per electronic health record review.
Time Frame: Up to 6 months after cancer diagnosis date
Population: Subjects who received a referral for cancer treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Mailed FIT Intervention - Age Group 50-75 | Trial Usual Care - Age Group 50-75
Number analyzed (Participants) | 5 | 2
Participants | 4 | 2

7. Secondary Outcome: Number of Subjects Mailed FITs Completed After Two Rounds of Annual FIT Outreach
Description: "Number of annual FIT screenings completed (0, 1, or 2) by subjects who received Intervention (Age Group 50-75) after two annual rounds of mailed FIT outreach per electronic health record review.
Time Frame: Round 1 time frame: at 6 months after randomization; Round 2 time frame: at 6 months after determining eligibility for Round 2
Population: Subjects who are 50-75 years old received study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Completed 0 Annual FITs: Completed 0 Annual FITs
- Completed 1 Annual FIT Screening Only in Year 1: Completed 1 Annual FIT Screening Only in Year 1
- Completed 1 Annual FIT Screening Only in Year 2: Completed 1 Annual FIT Screening Only in Year 2
- Completed 2 Annual FIT Screenings in Year 1 and Year 2: Completed 2 Annual FIT Screenings in Year 1 and Year 2
Arm/Group | Completed 0 Annual FITs | Completed 1 Annual FIT Screening Only in Year 1 | Completed 1 Annual FIT Screening Only in Year 2 | Completed 2 Annual FIT Screenings in Year 1 and Year 2
Number analyzed (Participants) | 2001 | 2001 | 1624 | 1624
Participants | 1372 | 261 | 116 | 252

8. Secondary Outcome: Incremental Cost of Each Additional Patient Screened in the Intervention Arm Compared to Usual Care (Trial - Age Group 50-75)
Description: Comparison of the programmatic costs incurred and number of subjects screened in Arm 1(Trial Mailed FIT Intervention - Age Group 50-75) compared to Arm 2 (Trial Usual Care - Age Group 50-75), measured as cost of intervention minus the cost of usual care, divided by the number screened in Arm 1 minus the number screened in Arm 2. Intervention costs will be assessed using periodic episodes of direct observation of mailed FIT outreach activities, time logs maintained by the intervention team, and assembly of administrative data capturing non-personnel/non-labor expenditures, such as costs associated with materials printing, FIT processing, and mailing costs. Usual care costs will be assessed using a combination of clinic observations and interviews with staff.
Time Frame: Through study completion, up to 36 months after randomization
Reporting Status: Not Posted

9. Secondary Outcome: The Proportion of Subjects, Ages 45-49, Who Are Current With CRC Screening
Description: The proportion of subjects in Arm 3 (Sub-study Mailed FIT Intervention Enhanced Envelope - Age Group 45-49) and Arm 4 (Sub-study Mailed FIT Active Comparator Envelope - Age Group 45-49) who are current with any CRC screening compared to baseline, using any of the screening modalities recommended by the United States Preventive Services Task Force (FIT, fecal occult blood test [FOBT], FIT-DNA, colonoscopy, flexible sigmoidoscopy, flexible sigmoidoscopy with FIT, CT colonography) per electronic health record review.
Time Frame: Up to 6 months after randomization
Population: Screening-eligible population, aged 45-49 years old.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Mailed FIT Intervention Enhanced Envelope - Age Group 45-49 Enhanced Envelope: Subjects randomized to this arm are 45-49 years of age and eligible for CRC screening using FIT per electronic health record at one FQHC. This arm receives a mailed FIT in an enhanced mailing envelope and up to two reminder letters.
- Active Comparator: Sub-study Mailed FIT Comparator Plain Envelope - Age Group 45-49: Subjects randomized to this arm are 45-49 years of age and eligible for CRC screening using FIT per electronic health record at one FQHC. This arm receives a mailed FIT in a plain envelope and up to two reminder letters.
Arm/Group | Experimental: Mailed FIT Intervention Enhanced Envelope - Age Group 45-49 Enhanced Envelope | Active Comparator: Sub-study Mailed FIT Comparator Plain Envelope - Age Group 45-49
Number analyzed (Participants) | 158 | 158
Participants
  Screening-eligible population, aged 45-49 years old | 158 | 158
  Count of screened participants | 53 | 45

10. Secondary Outcome: Proportion of Subjects, Ages 45-49, Who Completed Mailed FIT at 60 Days
Description: The proportion of subjects in Arm 3 (Intervention Enhanced Envelope - Age Group 45-49) compared to subjects in Arm 4 (Intervention Active Comparator Envelope - Age Group 45-49) who returned a completed FIT.
Time Frame: 60 days after randomization
Population: Subjects who are between 45-49 old completed mailed FIT at 60 days
Measure: Count of Participants; unit: Participants
Groups:
- Trial Mailed FIT Intervention - Age Group 45-49: Subjects randomized to this arm are 45-49 years of age and eligible for CRC screening using FIT per electronic health record at one site.
  Trial Mailed FIT Intervention - Age Group 45- 49: Subjects are mailed an introductory letter advising them that they will receive an FIT kit in the mail. Next, subjects are mailed a FIT packet in an envelope that contains a cover letter, CRC information sheet, FIT instruction sheet, and FIT kit with a pre-paid return envelope. Subjects receive up to two mailed letters reminding them to complete and return the FIT. Subjects receive FIT results via letter or phone call.
- Trial Usual Care - Age Group 45-49: Subjects randomized to this arm are 45-49 years of age and eligible for CRC screening using FIT per electronic health record at one site.
Arm/Group | Trial Mailed FIT Intervention - Age Group 45-49 | Trial Usual Care - Age Group 45-49
Number analyzed (Participants) | 158 | 158
Participants | 34 | 20

11. Secondary Outcome: Proportion of Subjects Who Completed a Follow up (Diagnostic) Colonoscopy
Description: The proportion of subjects in Arm 3 (Sub-study Mailed FIT Intervention Enhanced Envelope - Age Group 45-49) and Arm 4 (Sub-study Mailed FIT Active Comparator Plain Envelope - Age Group 45-40) with a positive (abnormal) FIT/FOBT result for whom colonoscopy is deemed to be clinically appropriate by the subject's provider who completes a follow-up (diagnostic) colonoscopy per electronic health record review.
Time Frame: Up to 6 months after abnormal FIT result date
Population: Subjects who are 45-49 years old completed study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Mailed FIT Intervention - Age Group 45-49 | Trial Usual Care - Age Group 45-49
Number analyzed (Participants) | 158 | 158
Participants
  positive (abnormal) FIT/FOBT result | 2 | 1
  completed a follow-up colonoscopy | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: This study does not require adverse event collection. Adverse events and mortality data were not collected.
Groups:
- Experimental: Trial Mailed FIT - Age Group 50-75: Subjects randomized to this arm are 50-75 years of age and eligible for colorectal cancer screening using FIT per electronic health record at either of the two study sites. This arm receives a mailed FIT and up to two reminder letters.
- No Intervention: Trial Usual Care - Age Group 50-75: Subjects randomized to this arm are 50-75 years of age and eligible for colorectal cancer screening using FIT per electronic health record at either of the two study sites. This arm receives the usual care.
- Experimental: Sub-study Mailed FIT Age Group 45-49 Enhanced Envelope: Subjects randomized to this arm are 45-49 years of age and eligible for colorectal cancer screening using FIT per electronic health record at one study site. This arm receives a mailed FIT in an enhanced mailing envelope and up to two reminder letters.
- Active Comparator: Sub-study Mailed FIT Comparator Plain Envelope - Age Group 45-49: Subjects randomized to this arm are 45-49 years of age and eligible for colorectal cancer screening using FIT per electronic health record at one study site. This arm receives a mailed FIT in a plain envelope and up to two reminder letters.
Arm/Group | Experimental: Trial Mailed FIT - Age Group 50-75 | No Intervention: Trial Usual Care - Age Group 50-75 | Experimental: Sub-study Mailed FIT Age Group 45-49 Enhanced Envelope | Active Comparator: Sub-study Mailed FIT Comparator Plain Envelope - Age Group 45-49
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT04406714/Prot_SAP_000.pdf